CLINICAL TRIAL: NCT03649412
Title: A Two Part, Non-randomised, Open Label Study Designed to Assess the Pharmacokinetic Profile of Modified Release Prototype Coated Tablet Formulations of GSK2982772 Relative to an Immediate Release Reference Tablet Formulation at a Fixed Strength (Part A) and the Pharmacokinetic Profile of Alternative Tablet Strengths of the Selected Modified Release Prototype Coated Tablet Formulation (Part B, Optional) in Healthy Participants
Brief Title: A Study to Investigate the Pharmacokinetics (PK) of Modified Release (MR) Prototype Coated Tablet Formulations of GSK2982772
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 209261; 2018-002370-48 (EudraCT Number)
Record Dates: First submitted 2018-08-24; First posted 2018-08-28 (Actual); Results first posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Autoimmune Diseases
Keywords: Tablet formulation; Sequence; Immediate release; Pharmacokinetic
MeSH Terms: conditions — Autoimmune Diseases | interventions — GSK2982772

STUDY DESIGN:
Intervention Model Description: Part A will be a 6-period, 6-way fixed sequence design, in which up to 4 MR tablet prototype coated formulation will be evaluated, following single dose administration (240 mg) in fasted or fed state. There will be a minimum 7-day washout between doses. Part B of the study is optional. Following the final period of Part A, there will be an interim review to determine whether to proceed with optional Part B, and if so, the formulations and tablet strengths to be investigated in Part B. The Part B of the study will be a 7-period fixed sequence which will evaluate the selected MR prototype coated tablet formulation(s) at different tablet strengths or as multiple unit doses.
Masking Description: There will be no masking as this is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects in Part A (Experimental): Subjects in Part A will receive GSK2982772 MR (Period 1, 3, 4, 5 and 6) and GSK2982772 IR (Period 2).
  Interventions: Drug: GSK2982772 Modified Release; Drug: GSK2982772 Immediate Release
- Subjects in Part B (Experimental): Subjects in Part B will receive GSK2982772 MR.
  Interventions: Drug: GSK2982772 Modified Release

INTERVENTIONS:
Drug: GSK2982772 Modified Release — GSK2982772 MR will be available as MR prototype coated tablet with unit dose strength of 240 mg in Part A. In Part B, GSK2982772 MR prototype coated tablet with unit dose strength of 120 mg (may be changed following interim review of Part B) will be administered by subjects. GSK2982772 MR will be administered orally with 240 milliliter (mL) of water.
Drug: GSK2982772 Immediate Release — In part A, GSK2982772 IR tablet will be available with unit dose strength of 30 mg and the total dose administered by subjects will be 240 mg (8 tablets of dose strength 30 mg) orally with 240 mL of water
  Arms: Subjects in Part A

SUMMARY:
Previous clinical studies of immediate release (IR) formulations of GSK2982772 resulted in a high peak to trough ratio of GSK2982772. Additionally, the short half-life for GSK2982772 (approximately 2 to 3 hours) necessitates twice a daily (BID) or thrice daily (TID) dosing of an IR formulation. As a result, MR formulations using a polymer matrix approach with minitablets in capsule and MR tablet formulations were investigated. The emerging PK data of the MR formulations investigated to date have demonstrated that a once daily (QD) PK profile can be achieved in the fasted state but the polymer matrix formulation is susceptible to food effects when administered with a high fat breakfast. The purpose of this study is to evaluate MR prototype coated tablet formulations. This study will evaluate the PK of MR prototype coated tablet formulations of GSK2982772. The study is divided into two parts; Part A and Part B. The MR tablet coating used in Part A and the initial periods of Part B will have an aperture drilled into the enteric coating of either side of the tablet. This allows some drug release to commence in the stomach whilst providing controlled release throughout the gastrointestinal (GI) tract. In Part B only, a new investigational medicinal product (IMP) will be manufactured to allow comparison of the tablet coating either with apertures (i.e., drilled) or without apertures (i.e., full coat/non drilled). Part A will be a 6-period, 6-way fixed sequence design, up to 4 MR tablet prototype coated formulations will be evaluated in fasted state at 240 milligrams (mg). Periods 1, 2 and 3 will evaluate MR1, IR tablet and MR2 respectively. Periods 4, 5 and 6 will be flexible and the dosing regimen will be dependent on the outcome of Periods 1 to 3. In addition, the impact of food (high fat meal, standard breakfast or administration 30 or 60 minutes before a standard breakfast) on selected MR prototype coated tablet formulations may also be evaluated in Period 4, 5 or 6 of Part A. Each inpatient period for MR regimens (Periods 1, 3, 4 to 6) will consist of 4 days and 3 nights, and the inpatient period for the IR tablet (Period 2) will consist of 3 days and 2 nights. There will be a minimum washout of 7 days between doses, and a follow-up visit will occur at 7 to 9 days after the last study treatment. The Part B of the study will be a 7-period fixed sequence which will evaluate the selected MR prototype coated tablet formulation(s) at different tablet strengths or as multiple unit doses and with or without apertures in the tablet coatings. There will be an interim review after each period 1 to 5 of Part B to select the dose level, formulation and prandial status for each subsequent period. An interim data review after Part B Period 6 will determine if optional Period 7 is required and the dose level, dosing time (morning or evening), formulation and prandial status for that period. Each inpatient period will consist of a 4-day and 3-night with a minimum of 7 days washout between doses. A follow-up visit will occur at 7 to 9 days after the last study treatment. Approximately 33 subjects will be enrolled in the study. The total duration for Part A will be approximately 10-12 weeks and 10-14 weeks for Part B (including screening period of approximately 4 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Subject at the time of participation must be 18 to 65 years of age.
* Subjects who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Body weight greater than or equal to 50 kilogram (kg) and body mass index within the range 19.0 to 32.0 kg per squared meter (kg/m^2) (inclusive).
* Male or female subjects where male subjects are eligible to participate if they agree to the following during the intervention period until completion of the final follow up visit after the last dose of study treatment; refrain from sperm donation; plus either be abstinent from heterosexual or homosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent; or must agree to use contraception/barrier like use a male condom and should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak when having sexual intercourse with a woman of childbearing potential who is not currently pregnant; agree to use male condom when engaging in any activity that allows for passage of ejaculate to another person.
* The eligible female subjects can participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: is not a woman of childbearing potential (WOCBP); is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of less than 1 percentage per year), preferably with low user dependency, for at least 30 days before first dose until completion of the final follow up visit after the last dose of study treatment and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction from Day 1 until 3 months after the last dose. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention; a WOCBP must have a negative highly sensitive serum pregnancy test within 24 hours before the first dose of study intervention; additional requirements for pregnancy testing during and after study intervention must be followed; the investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* Capable of giving an Informed Consent.

Exclusion Criteria:

* History of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal (GI), endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data.
* Any history of suicidal behavior within the past 6 months or any history of attempted suicide in subject's lifetime.
* History of clinically significant psychiatric disorders as judged by the investigator. Depression requiring treatment in the last 2 years.
* History of herpes zoster (shingles) reactivation.
* History or diagnosis of obstructive Sleep Apnea.
* History of a significant respiratory disorder. Childhood asthma that has fully resolved is permitted.
* History or current evidence of febrile seizures, epilepsy, convulsions, significant head injury, or other significant neurologic conditions.
* A positive diagnostic tuberculosis (TB) test at screening defined as a positive QuantiFERON-TB Gold test or T-spot test. In cases where the QuantiFERON or T-spot test is indeterminate, the subject may have the test repeated once, but they will not be eligible for the study unless the second test is negative.
* History of GI surgery (with exception of appendectomy).
* History of cholecystectomy or gall stones.
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever is allowed unless it is active.
* Alanine transaminase (ALT) greater than 1.5 times upper limit of normal (ULN).
* Bilirubin greater than 1.5 times ULN (isolated bilirubin greater than 1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35 percentage of total).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome).
* Corrected QT interval (QTcF) greater than 450 milliseconds (msec).
* Past or intended use of over-the-counter or prescription medication including herbal medications within 7 days prior to dosing (paracetamol/acetaminophen [up to 2 gram per day], hormone replacement therapy and hormonal contraception are permitted).
* Live or attenuated vaccine(s) within 30 days of enrolment, or plans to receive such vaccines during the study or plans to receive a vaccine within 30 days plus 5 half lives, of the last dose of study medication.
* Participation in the study would result in loss of blood or blood products in excess of 500 mL within a 56 day period; therefore donation or loss of greater than 400 mL of blood within the previous 3 months.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Current enrolment or past participation within the last 3 months before signing of consent in this or any other clinical study involving an investigational study treatment or any other type of medical research.
* Subjects who have previously been enrolled in this study. Subjects in Part A of this study are not permitted to participate in Part B.
* Current or history of renal disease or estimated glomerular filtration rate by chronic kidney disease epidemiology collaboration (CKD-EPI) equation calculation less than 60 milliliter (mL) per minute per 1.73 m^2 at screening.
* Presence of Hepatitis B surface antigen (HBsAg) at screening. Positive Hepatitis C antibody test result at screening or within 3 months prior to first dose. As potential for and magnitude of immunosuppression with this compound is unknown, subjects with presence of Hepatitis B core antibody (HBcAb) should be excluded. Subjects positive for HBsAg and/or positive for anti-HBc antibody (regardless of anti-HBs antibody status) are excluded.
* An elevated C-reactive protein (CRP) outside the normal reference range.
* Confirmed positive pre-study drug/alcohol screen.
* Positive human immunodeficiency virus (HIV) antibody test.
* Regular use of known drugs of abuse, or history of drug or alcohol abuse in the past 5 years.
* Regular alcohol consumption within 6 months prior to the study defined as an average weekly intake of greater than 21 units for males or greater than14 units for females. One unit is equivalent to 8 gram of alcohol: a half-pint (approximately 240 mL) of beer or 1 (25 mL) measure of spirits, 1.5 to 2 units is 1 glass (125 mL) of wine, depending on type.
* Current use or history of regular use of tobacco- or nicotine-containing products within 6 months prior to screening. A carbon monoxide breath test reading of greater than 10 parts per million (ppm).
* Sensitivity to any of the study treatments, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.
* Subjects who do not have suitable veins for multiple venipuncture's/cannulation as assessed by the investigator at screening.
* Total cholesterol greater than or equal to 300 mg per deciliter (mg/dL) (greater than or equal to 7.77 millimole per liter [mmol]/L]) or triglycerides greater than or equal to 250 mg/dL (greater than or equal to 2.82 mmol/L).
* Subjects who are study site or sponsor employees, or immediate family members of a study site or sponsor employee.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available, within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided, after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided, for an initial period of 12 months but an extension can be granted, when justified for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Tompson D, Whitaker M, Pan R, Johnson G, Fuller T, Zann V, McKenzie L, Abbott-Banner K, Hawkins S, Powell M. Development of a Once-Daily Modified-Release Formulation for the Short Half-Life RIPK1 Inhibitor GSK2982772 using DiffCORE Technology. Pharm Res. 2022 Jan;39(1):153-165. doi: 10.1007/s11095-021-03124-7. Epub 2022 Jan 5. PMID 34988780

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, 2-part (Part A & B), single dose study in healthy participants to assess modified release (MR) prototype coated tablet formulations of GSK2982772 compared to an immediate release reference tablet formulation.
Pre-assignment Details: A total of 33 participants were enrolled in this study. In Part A, 16 participants were enrolled but 1 replacement participant was added (total=17). Participants from Part A did not continue to Part B. In Part B, 16 participants were enrolled.
Groups:
- MR 12h Fast/IR Fast/MR18h Fast/MR 18h Fed/MR 12h Fed/MR16hFast: Participants in Part A received a single dose of 240 milligrams (mg) GSK2982772 MR-12 hour (h) tablet (80 percent [%] release in 12 hours) in fasted (fast) state in Period 1 followed by a single dose of GSK2982772 240 mg (8x30mg) immediate release (IR) tablet in fasted state in Period 2 followed by a single dose of 240 mg GSK2982772 MR-18h (80% release in 18 hours) tablet in fasted state in Period 3. In Period 4, participants received a single dose of 240 mg GSK2982772 MR-18h tablet after a high-fat meal (fed state) followed by a single dose of MR-12h tablet after a high fat meal (fed state) in Period 5. In Period 6, participants received a single dose of 240 mg of GSK2982772 of MR-16h tablet (80% release in 16 hours) in a fasted state. There was a washout of 7 days between each treatment period. All doses were administered orally with 240 milliliters (mL) of water.
- MR 480Fast/960Fast/480Fed/120Fast/480 Fed (Ent)/480 Fed(Std): Participants in Part B received a single dose of 480 mg GSK2982772 MR-16h tablet (80% release in 16 hours) in a fasted state in Period 1 followed by a single dose 960 mg GSK2982772 MR-16h tablet in a fasted state in Period 2 followed by a single dose of 480 mg GSK2982772 MR-16h tablet after a high-fat meal (fed state) in Period 3. In Period 4, participants received a single dose of 120 mg GSK2982772 MR-16h tablet in a fasted state followed by a single dose of 480 mg GSK2982772 MR-16h enteric (Ent) coated tablet after a high-fat meal (fed state) in Period 5. In Period 6, participants received a single dose of 480 mg GSK2982772 MR-16h tablet after a standard meal (fed state).There was a washout of 7 days between each treatment period. All doses were administered orally with 240 mL of water.
Period: Part A, Period 1 (4 Days)
Arm/Group | MR 12h Fast/IR Fast/MR18h Fast/MR 18h Fed/MR 12h Fed/MR16hFast | MR 480Fast/960Fast/480Fed/120Fast/480 Fed (Ent)/480 Fed(Std)
Started | 16 | 0
Completed | 16 | 0
Not Completed | 0 | 0
Period: Part A, Washout Period 1 (7 Days)
Arm/Group | MR 12h Fast/IR Fast/MR18h Fast/MR 18h Fed/MR 12h Fed/MR16hFast | MR 480Fast/960Fast/480Fed/120Fast/480 Fed (Ent)/480 Fed(Std)
Started | 16 | 0
Completed | 15 | 0
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0
Period: Part A, Period 2 (3 Days)
Arm/Group | MR 12h Fast/IR Fast/MR18h Fast/MR 18h Fed/MR 12h Fed/MR16hFast | MR 480Fast/960Fast/480Fed/120Fast/480 Fed (Ent)/480 Fed(Std)
Started | 16 (1 Replacement par. was enrolled & dosed) | 0
Completed | 16 | 0
Not Completed | 0 | 0
Period: Part A, Washout Period 2 (7 Days)
Arm/Group | MR 12h Fast/IR Fast/MR18h Fast/MR 18h Fed/MR 12h Fed/MR16hFast | MR 480Fast/960Fast/480Fed/120Fast/480 Fed (Ent)/480 Fed(Std)
Started | 16 | 0
Completed | 16 | 0
Not Completed | 0 | 0
Period: Part A, Period 3 (4 Days)
Arm/Group | MR 12h Fast/IR Fast/MR18h Fast/MR 18h Fed/MR 12h Fed/MR16hFast | MR 480Fast/960Fast/480Fed/120Fast/480 Fed (Ent)/480 Fed(Std)
Started | 16 | 0
Completed | 16 | 0
Not Completed | 0 | 0
Period: Part A, Washout Period 3 (7 Days)
Arm/Group | MR 12h Fast/IR Fast/MR18h Fast/MR 18h Fed/MR 12h Fed/MR16hFast | MR 480Fast/960Fast/480Fed/120Fast/480 Fed (Ent)/480 Fed(Std)
Started | 16 | 0
Completed | 16 | 0
Not Completed | 0 | 0
Period: Part A, Period 4 (4 Days)
Arm/Group | MR 12h Fast/IR Fast/MR18h Fast/MR 18h Fed/MR 12h Fed/MR16hFast | MR 480Fast/960Fast/480Fed/120Fast/480 Fed (Ent)/480 Fed(Std)
Started | 16 | 0
Completed | 16 | 0
Not Completed | 0 | 0
Period: Part A, Washout Period 4 (7 Days)
Arm/Group | MR 12h Fast/IR Fast/MR18h Fast/MR 18h Fed/MR 12h Fed/MR16hFast | MR 480Fast/960Fast/480Fed/120Fast/480 Fed (Ent)/480 Fed(Std)
Started | 16 | 0
Completed | 14 | 0
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Part A, Period 5 (4 Days)
Arm/Group | MR 12h Fast/IR Fast/MR18h Fast/MR 18h Fed/MR 12h Fed/MR16hFast | MR 480Fast/960Fast/480Fed/120Fast/480 Fed (Ent)/480 Fed(Std)
Started | 12 (Two participant did not start in Period 5) | 0
Completed | 12 | 0
Not Completed | 0 | 0
Period: Part A, Washout Period 5 (7 Days)
Arm/Group | MR 12h Fast/IR Fast/MR18h Fast/MR 18h Fed/MR 12h Fed/MR16hFast | MR 480Fast/960Fast/480Fed/120Fast/480 Fed (Ent)/480 Fed(Std)
Started | 12 | 0
Completed | 11 | 0
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Part A, Period 6 (4 Days)
Arm/Group | MR 12h Fast/IR Fast/MR18h Fast/MR 18h Fed/MR 12h Fed/MR16hFast | MR 480Fast/960Fast/480Fed/120Fast/480 Fed (Ent)/480 Fed(Std)
Started | 12 (1 of the participant who did not start Period 5 directly joined into Period 6) | 0
Completed | 12 | 0
Not Completed | 0 | 0
Period: Part B, Period 1 (4 Days)
Arm/Group | MR 12h Fast/IR Fast/MR18h Fast/MR 18h Fed/MR 12h Fed/MR16hFast | MR 480Fast/960Fast/480Fed/120Fast/480 Fed (Ent)/480 Fed(Std)
Started | 0 (Participants in Part A did not enter Part B) | 16 (16 new participants enrolled in Part B)
Completed | 0 | 16
Not Completed | 0 | 0
Period: Part B, Washout Period 1 (7 Days)
Arm/Group | MR 12h Fast/IR Fast/MR18h Fast/MR 18h Fed/MR 12h Fed/MR16hFast | MR 480Fast/960Fast/480Fed/120Fast/480 Fed (Ent)/480 Fed(Std)
Started | 0 | 16
Completed | 0 | 15
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Part B, Period 2 (4 Days)
Arm/Group | MR 12h Fast/IR Fast/MR18h Fast/MR 18h Fed/MR 12h Fed/MR16hFast | MR 480Fast/960Fast/480Fed/120Fast/480 Fed (Ent)/480 Fed(Std)
Started | 0 | 15
Completed | 0 | 15
Not Completed | 0 | 0
Period: Part B, Washout Period 2 (7 Days)
Arm/Group | MR 12h Fast/IR Fast/MR18h Fast/MR 18h Fed/MR 12h Fed/MR16hFast | MR 480Fast/960Fast/480Fed/120Fast/480 Fed (Ent)/480 Fed(Std)
Started | 0 | 15
Completed | 0 | 15
Not Completed | 0 | 0
Period: Part B, Period 3 (4 Days)
Arm/Group | MR 12h Fast/IR Fast/MR18h Fast/MR 18h Fed/MR 12h Fed/MR16hFast | MR 480Fast/960Fast/480Fed/120Fast/480 Fed (Ent)/480 Fed(Std)
Started | 0 | 15
Completed | 0 | 15
Not Completed | 0 | 0
Period: Part B, Washout Period 3 (7 Days)
Arm/Group | MR 12h Fast/IR Fast/MR18h Fast/MR 18h Fed/MR 12h Fed/MR16hFast | MR 480Fast/960Fast/480Fed/120Fast/480 Fed (Ent)/480 Fed(Std)
Started | 0 | 15
Completed | 0 | 15
Not Completed | 0 | 0
Period: Part B, Period 4 (4 Days)
Arm/Group | MR 12h Fast/IR Fast/MR18h Fast/MR 18h Fed/MR 12h Fed/MR16hFast | MR 480Fast/960Fast/480Fed/120Fast/480 Fed (Ent)/480 Fed(Std)
Started | 0 | 15
Completed | 0 | 15
Not Completed | 0 | 0
Period: Part B, Washout Period 4 (7 Days)
Arm/Group | MR 12h Fast/IR Fast/MR18h Fast/MR 18h Fed/MR 12h Fed/MR16hFast | MR 480Fast/960Fast/480Fed/120Fast/480 Fed (Ent)/480 Fed(Std)
Started | 0 | 15
Completed | 0 | 15
Not Completed | 0 | 0
Period: Part B, Period 5 (4 Days)
Arm/Group | MR 12h Fast/IR Fast/MR18h Fast/MR 18h Fed/MR 12h Fed/MR16hFast | MR 480Fast/960Fast/480Fed/120Fast/480 Fed (Ent)/480 Fed(Std)
Started | 0 | 14 (One participant did not start in Period 5)
Completed | 0 | 14
Not Completed | 0 | 0
Period: Part B, Washout Period 5 (7 Days)
Arm/Group | MR 12h Fast/IR Fast/MR18h Fast/MR 18h Fed/MR 12h Fed/MR16hFast | MR 480Fast/960Fast/480Fed/120Fast/480 Fed (Ent)/480 Fed(Std)
Started | 0 | 14
Completed | 0 | 13
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Part B, Period 6 (4days)
Arm/Group | MR 12h Fast/IR Fast/MR18h Fast/MR 18h Fed/MR 12h Fed/MR16hFast | MR 480Fast/960Fast/480Fed/120Fast/480 Fed (Ent)/480 Fed(Std)
Started | 0 | 14 (Participant who did not start Period 5 directly joined into Period 6)
Completed | 0 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MR 12h Fast/IR Fast/MR18h Fast/MR 18h Fed/MR 12h Fed/MR16hFast | MR 480Fast/960Fast/480Fed/120Fast/480 Fed (Ent)/480 Fed(Std) | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.5 (12.17) | 54.0 (6.30) | 48.6 (11.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 10 | 10 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ARABIC/NORTH AFRICAN HERITAGE | 1 | 0 | 1
  WHITE/CAUCASIAN/EUROPEAN HERITAGE | 16 | 13 | 29
  AFRICAN AMERICAN/AFRICAN HERITAGE | 0 | 1 | 1
  CENTRAL/SOUTH ASIAN HERITAGE | 0 | 1 | 1
  MULTIPLE | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part A: Area Under the Curve From Time Zero to Infinity (AUC[0-inf]) of GSK2982772 240 mg in IR Formulation
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis. PK parameters were analyzed using standard non-compartmental analysis. Participants in the 'Safety Population (all participants who received at least one dose of study treatment)' for whom a PK sample was obtained and analyzed were part of PK Population.
Time Frame: Pre-dose, 0.33, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Groups:
- Part A: IR 240 mg Fasted: Participants received a single oral dose of 240 mg (8x30mg) GSK2982772 IR tablet in a fasted state
Arm/Group | Part A: IR 240 mg Fasted
Number analyzed (Participants) | 16
Hours*microgram per milliliter | 14.355 (31.1)

2. Primary Outcome: Part A: AUC(0-inf) of GSK2982772 240 mg in MR Coated Tablet Formulation
Description: Blood samples were collected from participants at indicated time points for PK analysis. PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 36 and 48 hours post-dose
Population: PK Population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Groups:
- Part A: MR-12h 240 mg Fasted: Participants received a single oral dose of 240 mg GSK2982772 MR-12h tablet in fasted state
- Part A: MR-18h 240 mg Fasted: Participants received a single oral dose of 240 mg GSK2982772 MR-18h tablet in fasted state
- Part A: MR-16h 240 mg Fasted: Participants received a single oral dose of 240 mg GSK2982772 MR-16h tablet in fasted state
Arm/Group | Part A: MR-12h 240 mg Fasted | Part A: MR-18h 240 mg Fasted | Part A: MR-16h 240 mg Fasted
Number analyzed (Participants) | 12 | 13 | 7
Hours*microgram per milliliter | 7.757 (19.1) | 8.346 (27.7) | 7.080 (46.8)

3. Primary Outcome: Part A: AUC(0-inf) of GSK2982772 240 mg in MR Coated Tablet Formulation After High-fat Breakfast
Description: as for outcome 2
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 36 and 48 hours post-dose
Population: PK Population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Groups:
- Part A: MR-12h 240 mg Fed (High-Fat): Participants received a single oral dose of 240 mg GSK2982772 MR-12h tablet after a high fat meal in fed state
- Part A: MR-18h 240 mg Fed (High-fat): Participants received a single oral dose of 240 mg GSK2982772 MR-18h tablet after high fat meal in fed state
Arm/Group | Part A: MR-12h 240 mg Fed (High-Fat) | Part A: MR-18h 240 mg Fed (High-fat)
Number analyzed (Participants) | 7 | 12
Hours*microgram per milliliter | 9.372 (21.8) | 8.220 (37.2)

4. Primary Outcome: Part A: Area Under the Curve From Time Zero to the Last Measurable Concentration (AUC[0-t]) of GSK2982772 240 mg for IR Formulation
Description: Blood samples were collected from participants at indicated time points and analyzed for AUC (0-t). PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Pre-dose, 0.33, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part A: IR 240 mg Fasted
Number analyzed (Participants) | 16
Hours*microgram per milliliter | 14.269 (31.2)

5. Primary Outcome: Part A: AUC(0-t) of GSK2982772 240 mg for MR Coated Tablet Formulation
Description: as for outcome 4
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 36 and 48 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part A: MR-12h 240 mg Fasted | Part A: MR-18h 240 mg Fasted | Part A: MR-16h 240 mg Fasted
Number analyzed (Participants) | 16 | 16 | 12
Hours*microgram per milliliter | 8.175 (23.9) | 7.828 (28.5) | 7.365 (36.4)

6. Primary Outcome: Part A: AUC(0-t) of GSK2982772 240 mg for MR Coated Tablet Formulation After High-fat Breakfast
Description: as for outcome 4
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 36 and 48 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part A: MR-12h 240 mg Fed (High-Fat) | Part A: MR-18h 240 mg Fed (High-fat)
Number analyzed (Participants) | 12 | 16
Hours*microgram per milliliter | 9.359 (23.1) | 8.384 (32.7)

7. Primary Outcome: Part A: Area Under the Curve From Time Zero to 24 Hours (AUC[0-24]) of GSK2982772 240 mg for IR Formulation
Description: Blood samples were collected from participants at indicated time points and analyzed for AUC (0-24). PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Pre-dose, 0.33, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part A: IR 240 mg Fasted
Number analyzed (Participants) | 16
Hours*microgram per milliliter | 14.268 (31.2)

8. Primary Outcome: Part A: AUC(0-24) of GSK2982772 240 mg for MR Coated Tablet Formulation
Description: as for outcome 7
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part A: MR-12h 240 mg Fasted | Part A: MR-18h 240 mg Fasted | Part A: MR-16h 240 mg Fasted
Number analyzed (Participants) | 16 | 16 | 12
Hours*microgram per milliliter | 6.670 (24.9) | 5.784 (31.8) | 5.466 (33.1)

9. Primary Outcome: Part A: AUC(0-24) of GSK2982772 240 mg for MR Coated Tablet Formulation After High-fat Breakfast
Description: as for outcome 7
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Groups:
- Part A: MR-12h 240mg Fed (High-Fat): Participants received a single oral dose of 240 mg GSK2982772 MR-12h tablet after a high fat meal in fed state
Arm/Group | Part A: MR-12h 240mg Fed (High-Fat) | Part A: MR-18h 240 mg Fed (High-fat)
Number analyzed (Participants) | 12 | 16
Hours*microgram per milliliter | 7.136 (33.5) | 5.821 (32.1)

10. Primary Outcome: Part A: Maximum Observed Concentration (Cmax) of GSK2982772 240 mg for IR Formulation
Description: Blood samples were collected from participants at indicated time points and analyzed for Cmax. PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Pre-dose, 0.33, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part A: IR 240 mg Fasted
Number analyzed (Participants) | 16
Microgram per milliliter | 3.177 (40.1)

11. Primary Outcome: Part A: Cmax of GSK2982772 240 mg for MR Coated Tablet Formulation
Description: as for outcome 10
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 36 and 48 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part A: MR-12h 240 mg Fasted | Part A: MR-18h 240 mg Fasted | Part A: MR-16h 240 mg Fasted
Number analyzed (Participants) | 16 | 16 | 12
Microgram per milliliter | 0.682 (39.4) | 0.527 (24.4) | 0.466 (27.5)

12. Primary Outcome: Part A: Cmax of GSK2982772 240 mg for MR Coated Tablet Formulation After High-fat Breakfast
Description: as for outcome 10
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 36 and 48 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part A: MR-12h 240 mg Fed (High-Fat) | Part A: MR-18h 240 mg Fed (High-fat)
Number analyzed (Participants) | 12 | 16
Microgram per milliliter | 0.824 (47.5) | 0.678 (47.0)

13. Primary Outcome: Part A: Concentration at 24 Hours Post-dose (C24h) of GSK2982772 240 mg for IR Formulation
Description: Blood samples were collected from participants at indicated time points and analyzed for C24h. PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part A: IR 240 mg Fasted
Number analyzed (Participants) | 16
Microgram per milliliter | 0.015 (60.8)

14. Primary Outcome: Part A: C24h of GSK2982772 240 mg for MR Coated Tablet Formulation
Description: as for outcome 13
Time Frame: 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part A: MR-12h 240 mg Fasted | Part A: MR-18h 240 mg Fasted | Part A: MR-16h 240 mg Fasted
Number analyzed (Participants) | 16 | 16 | 12
Microgram per milliliter | 0.196 (64.8) | 0.211 (63.1) | 0.165 (98.3)

15. Primary Outcome: Part A: C24h of GSK2982772 240 mg for MR Coated Tablet Formulation After High-fat Breakfast
Description: as for outcome 13
Time Frame: 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part A: MR-12h 240 mg Fed (High-Fat) | Part A: MR-18h 240 mg Fed (High-fat)
Number analyzed (Participants) | 12 | 16
Microgram per milliliter | 0.213 (70.4) | 0.265 (85.5)

16. Primary Outcome: Part A: Time to Cmax (Tmax) of GSK2982772 240 mg for IR Formulation
Description: Blood samples were collected from participants at indicated time points and analyzed for Tmax. PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Pre-dose, 0.33, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: IR 240 mg Fasted
Number analyzed (Participants) | 16
Hours | 2.000 [1.00 to 5.00]

17. Primary Outcome: Part A: Tmax of GSK2982772 240 mg for MR Coated Tablet Formulation
Description: as for outcome 16
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 36 and 48 hours post-dose
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: MR-12h 240 mg Fasted | Part A: MR-18h 240 mg Fasted | Part A: MR-16h 240 mg Fasted
Number analyzed (Participants) | 16 | 16 | 12
Hours | 5.000 [4.00 to 12.03] | 10.000 [4.00 to 24.20] | 6.000 [4.00 to 16.00]

18. Primary Outcome: Part A: Tmax of GSK2982772 240 mg for MR Coated Tablet Formulation After High-fat Breakfast
Description: as for outcome 16
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 36 and 48 hours post-dose
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: MR-12h 240 mg Fed (High-Fat) | Part A: MR-18h 240 mg Fed (High-fat)
Number analyzed (Participants) | 12 | 16
Hours | 8.000 [2.00 to 22.00] | 11.000 [8.00 to 22.32]

19. Primary Outcome: Part A: Terminal Half-life (t1/2) of GSK2982772 240 mg for IR Formulation
Description: Blood samples were collected from participants at indicated time points and analyzed for t1/2. PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Pre-dose, 0.33, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part A: IR 240 mg Fasted
Number analyzed (Participants) | 16
Hours | 3.288 (0.5010)

20. Primary Outcome: Part A: t1/2 of GSK2982772 240 mg for MR Coated Tablet Formulation
Description: as for outcome 19
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 36 and 48 hours
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part A: MR-12h 240 mg Fasted | Part A: MR-18h 240 mg Fasted | Part A: MR-16h 240 mg Fasted
Number analyzed (Participants) | 16 | 16 | 12
Hours | 6.329 (2.1447) | 6.953 (2.4983) | 7.532 (2.2685)

21. Primary Outcome: Part A: t1/2 of GSK2982772 240 mg for MR Coated Tablet Formulation After High-fat Breakfast
Description: as for outcome 19
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 36 and 48 hours
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part A: MR-12h 240mg Fed (High-Fat) | Part A: MR-18h 240 mg Fed (High-fat)
Number analyzed (Participants) | 12 | 16
Hours | 7.763 (1.4693) | 6.589 (1.0499)

22. Primary Outcome: Part B: AUC(0-inf) of GSK2982772 for MR Coated Tablet Formulation After a High Fat Breakfast
Description: Blood samples were collected from participants at indicated time points and analyzed for AUC(0-inf). PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 36 and 48 hours post-dose
Population: PK Population. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Groups:
- Part B: MR-16h 480mg Fed (High-Fat): Participants received a single oral dose of 480 mg GSK2982772 MR-16h (80% release in 16 hours) tablet after high fat breakfast (fed state)
- Part B: MR-16h 480mg Fed (High-Fat) (Enteric Coated): Participants received a single oral dose of 480 mg GSK2982772 MR-16h (80% release in 16 hours) enteric coated tablet after a high fat breakfast (fed state)
Arm/Group | Part B: MR-16h 480mg Fed (High-Fat) | Part B: MR-16h 480mg Fed (High-Fat) (Enteric Coated)
Number analyzed (Participants) | 11 | 8
Hours*microgram per milliliter | 20.121 (46.2) | 20.178 (62.8)

23. Primary Outcome: Part B: AUC(0-t) of GSK2982772 for MR Coated Tablet Formulation After a High Fat Breakfast
Description: Blood samples were collected from participants at indicated time points and analyzed for AUC(0-t). PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 36 and 48 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part B: MR-16h 480mg Fed (High-Fat) | Part B: MR-16h 480mg Fed (High-Fat) (Enteric Coated)
Number analyzed (Participants) | 15 | 14
Hours*microgram per milliliter | 19.865 (39.7) | 17.861 (47.1)

24. Primary Outcome: Part B: Cmax of GSK2982772 for MR Coated Tablet Formulation After a High Fat Breakfast
Description: as for outcome 10
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 36 and 48 hours post-dose post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part B: MR-16h 480mg Fed (High-Fat) | Part B: MR-16h 480mg Fed (High-Fat) (Enteric Coated)
Number analyzed (Participants) | 15 | 14
Hours*microgram per milliliter | 1.896 (63.3) | 1.791 (75.0)

25. Primary Outcome: Part B: C24h of GSK2982772 for MR Coated Tablet Formulation After a High Fat Breakfast
Description: as for outcome 13
Time Frame: 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part B: MR-16h 480mg Fed (High-Fat) | Part B: MR-16h 480mg Fed (High-Fat) (Enteric Coated)
Number analyzed (Participants) | 15 | 14
Microgram per milliliter | 0.622 (132.9) | 1.176 (80.6)

26. Primary Outcome: Part B: Tmax of GSK2982772 for MR Coated Tablet Formulation After a High Fat Breakfast
Description: as for outcome 16
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 36 and 48 hours post-dose
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part B: MR-16h 480mg Fed (High-Fat) | Part B: MR-16h 480mg Fed (High-Fat) (Enteric Coated)
Number analyzed (Participants) | 15 | 14
Hours | 12.000 [6.00 to 28.00] | 22.008 [10.00 to 24.05]

27. Primary Outcome: Part B: t1/2 of GSK2982772 for MR Coated Tablet Formulation After a High Fat Breakfast
Description: as for outcome 19
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 36 and 48 hours post-dose
Population: PK Population. Only those participants with data available at specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part B: MR-16h 480mg Fed (High-Fat) | Part B: MR-16h 480mg Fed (High-Fat) (Enteric Coated)
Number analyzed (Participants) | 11 | 8
Hours | 4.961 (1.0921) | 4.873 (1.9915)

28. Primary Outcome: Part A: Relative Bioavailability in Fed Versus Fasted Conditions (FrelFE) Based on AUC(0-inf) of GSK2982772 for MR Coated Tablet Formulation
Description: Blood samples were collected at indicated time points for analysis of FrelFE based on AUC of GSK2982772. Frel for AUC(0-inf) was calculated as Geometric mean of AUC(0-inf) of MR Fed/ Geometric mean of AUC(0-inf) of MR Fasted multiplied by 100.
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 36 and 48 hours post-dose
Population: PK Population. Only those participants with data available at specified time points were analyzed.
Measure: Number (90% Confidence Interval); unit: Percentage bioavailability
Groups:
- Part A: MR-18h 240mg Fed and MR-18h 240mg Fasted: Participants received a single oral dose of 240 mg GSK2982772 MR-18h (80% release in 18 hours) tablet in fed (high-fat) state and received MR-18h (80% release in 18 hours) tablet in fasted state
- Part A: MR-12h 240mg Fed and MR-12h 240mg Fasted: Participants received a single oral dose of 240 mg GSK2982772 MR-12h (80% release in 12 hours) tablet in fed (high-fat) state and received MR-12h (80% release in 12 hours) tablet in fasted state
Arm/Group | Part A: MR-18h 240mg Fed and MR-18h 240mg Fasted | Part A: MR-12h 240mg Fed and MR-12h 240mg Fasted
Number analyzed (Participants) | 13 | 12
Percentage bioavailability | 102.66 [88.84 to 118.63] | 113.66 [95.53 to 135.24]

29. Primary Outcome: Part A: FrelFE Based on AUC(0-t) of GSK2982772 for MR Coated Tablet Formulation
Description: Blood samples were collected at indicated time points for analysis of FrelFE based on AUC of GSK2982772. Frel for AUC(0-t) was calculated as Geometric mean of AUC(0-t) of MR Fed/Geometric mean of AUC(0-t) of MR Fasted multiplied by 100.
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 36 and 48 hours post-dose
Population: PK Population.
Measure: Number (90% Confidence Interval); unit: Percentage bioavailability
Arm/Group | Part A: MR-18h 240mg Fed and MR-18h 240mg Fasted | Part A: MR-12h 240mg Fed and MR-12h 240mg Fasted
Number analyzed (Participants) | 16 | 16
Percentage bioavailability | 107.11 [95.72 to 119.85] | 107.81 [95.16 to 122.14]

30. Primary Outcome: Part A: FrelFE Based on Cmax of GSK2982772 for MR Coated Tablet Formulation
Description: Blood samples were collected at indicated time points for analysis of FrelFE based on Cmax of GSK2982772. Frel for Cmax was calculated as Geometric mean of Cmax of MR Fed/Geometric mean of Cmax of MR Fasted multiplied by 100.
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 36 and 48 hours post-dose
Population: PK Population.
Measure: Number (90% Confidence Interval); unit: Percentage bioavailability
Arm/Group | Part A: MR-18h 240mg Fed and MR-18h 240mg Fasted | Part A: MR-12h 240mg Fed and MR-12h 240mg Fasted
Number analyzed (Participants) | 16 | 16
Percentage bioavailability | 128.79 [108.64 to 152.67] | 112.15 [92.90 to 135.38]

31. Primary Outcome: Part B: FrelFE of GSK2982772 Based on AUC(0-inf) for MR Coated Tablet Formulation in Fed vs Fasted State
Description: Blood samples were collected at indicated time points for analysis of FrelFE based on AUC(0-inf) of GSK2982772. Frel for AUC(0-inf) was calculated as Geometric mean of AUC(0-inf) of MR Fed/ Geometric mean of AUC(0-inf) of MR Fasted multiplied by 100.
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 36 and 48 hours post-dose
Population: PK Population. Only those participants with data available at specified time frame were analyzed.
Measure: Number (90% Confidence Interval); unit: Percentage bioavailability
Groups:
- Part B: MR-16h 480mg Fed (High-fat) and MR-16h 480mg Fasted: Participants received a single oral dose of 480 mg GSK2982772 MR-16h (80% release in 16 hours) tablet after high fat breakfast in fed state and received a single oral dose of 480 mg GSK2982772 MR-16 h (80% release in 16 hours) tablet in fasted state
- Part B: MR-16h 480mg Fed (Standard) and MR-16h 480mg Fasted: Participants received a single oral dose of 480 mg GSK2982772 MR-16h (80% release in 16 hours) tablet after a standard breakfast in fed state and received a single oral dose of 480mg GSK2982772 MR-16 h (80% release in 16 hours) tablet in fasted state
Arm/Group | Part B: MR-16h 480mg Fed (High-fat) and MR-16h 480mg Fasted | Part B: MR-16h 480mg Fed (Standard) and MR-16h 480mg Fasted
Number analyzed (Participants) | 11 | 12
Percentage bioavailability | 141.75 [113.47 to 177.07] | 97.13 [78.47 to 120.22]

32. Primary Outcome: Part B: FrelFE of GSK2982772 Based on AUC (0-t) for MR Coated Tablet Formulation in Fed vs Fasted State
Description: Blood samples were collected at indicated time points for analysis of FrelFE based on AUC (0-t) of GSK2982772. FrelFE for AUC (0-t) was calculated as Geometric mean of AUC (0-t) of MR Fed/ Geometric mean of AUC (0-t) of MR Fasted multiplied by 100.
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 36 and 48 hours post-dose
Population: PK Population.
Measure: Number (90% Confidence Interval); unit: Percentage bioavailability
Arm/Group | Part B: MR-16h 480mg Fed (High-fat) and MR-16h 480mg Fasted | Part B: MR-16h 480mg Fed (Standard) and MR-16h 480mg Fasted
Number analyzed (Participants) | 16 | 16
Percentage bioavailability | 129.63 [109.23 to 153.83] | 89.77 [75.37 to 106.92]

33. Primary Outcome: Part B: FrelFE of GSK2982772 Based on Cmax for MR Coated Tablet Formulation in Fed vs Fasted State
Description: Blood samples were collected at indicated time points for analysis of FrelFE based on Cmax of GSK2982772. FrelFE for Cmax was calculated as Geometric mean of Cmax of MR Fed/ Geometric mean of Cmax of MR Fasted multiplied by 100.
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 36 and 48 hours post-dose
Population: PK Population.
Measure: Number (90% Confidence Interval); unit: Percentage bioavailability
Groups:
- Part B: MR-16h 480mg Fed (High-fat) vs MR-16h 480mg Fasted: Participants received a single oral dose of 480 mg GSK2982772 MR-16h (80% release in 16 hours) tablet after high fat breakfast in fed state and received a single oral dose of 480 mg GSK2982772 MR-16 h (80% release in 16 hours) tablet in fasted state
Arm/Group | Part B: MR-16h 480mg Fed (High-fat) vs MR-16h 480mg Fasted | Part B: MR-16h 480mg Fed (Standard) and MR-16h 480mg Fasted
Number analyzed (Participants) | 16 | 16
Percentage bioavailability | 173.19 [138.68 to 216.28] | 102.39 [81.61 to 128.47]

34. Primary Outcome: Part B: Frel of GSK2982772 Based on AUC (0-inf) for MR Coated Tablet Formulation in Fasted State
Description: Blood samples were collected at indicated time points for analysis of Frel (dose) based on AUC (0-inf) of GSK2982772. Frel (dose) for AUC (0-inf) was calculated as Geometric mean of AUC (0-inf) of MR formulation (test dose) Fasted/ Geometric mean of AUC (0-inf) of MR Fasted formulation (reference dose) multiplied by 100.
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 36 and 48 hours post-dose
Population: PK Population. Only those participants with data available at specified time points were analyzed.
Measure: Number (90% Confidence Interval); unit: Percentage bioavailability
Groups:
- Part B: MR-16h 960mg Fasted and MR-16h 480mg Fasted: Participants received a single oral dose of 960 mg GSK2982772 MR-16h (80% release in 16 hours) tablet in fasted state and received 480 mg GSK2982772 MR-16 h (80% release in 16 hours) tablet in fasted state
- Part B: MR-16h 960mg Fasted vs MR-16h 120mg Fasted: Participants received a single oral dose of 960 mg GSK2982772 MR-16h (80% release in 16 hours) tablet in fasted state and received 120 mg GSK2982772 MR-16 h (80% release in 16 hours) tablet in fasted state
- Part B: MR-16h 480mg Fasted vs MR-16h 120mg Fasted: Participants received a single oral dose of 480 mg GSK2982772 MR-16h (80% release in 16 hours) tablet in fasted state and received 120 mg GSK2982772 MR-16 h (80% release in 16 hours) tablet in fasted state
Arm/Group | Part B: MR-16h 960mg Fasted and MR-16h 480mg Fasted | Part B: MR-16h 960mg Fasted vs MR-16h 120mg Fasted | Part B: MR-16h 480mg Fasted vs MR-16h 120mg Fasted
Number analyzed (Participants) | 10 | 14 | 14
Percentage bioavailability | 214.21 [171.24 to 267.95] | 530.86 [431.89 to 652.49] | 247.82 [201.70 to 304.49]

35. Primary Outcome: Part B: Frel of GSK2982772 Based on AUC (0-t) for MR Coated Tablet Formulation in Fasted State
Description: Blood samples were collected at indicated time points for analysis of Frel (dose) based on AUC(0-t) of GSK2982772. Frel (dose) for AUC(0-t) was calculated as Geometric mean of AUC(0-t) of MR formulation (test dose) Fasted/ Geometric mean of AUC(0-t) of MR Fasted formulation (reference dose) multiplied by 100.
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 36 and 48 hours post-dose
Population: PK Population.
Measure: Number (90% Confidence Interval); unit: Percentage bioavailability
Groups:
- Part B: MR-16h 960mg Fasted vs MR-16h 480mg Fasted: Participants received a single oral dose of 960 mg GSK2982772 MR-16h (80% release in 16 hours) tablet in fasted state and received 480 mg GSK2982772 MR-16 h (80% release in 16 hours) tablet in fasted state
Arm/Group | Part B: MR-16h 960mg Fasted vs MR-16h 480mg Fasted | Part B: MR-16h 960mg Fasted vs MR-16h 120mg Fasted | Part B: MR-16h 480mg Fasted vs MR-16h 120mg Fasted
Number analyzed (Participants) | 16 | 15 | 16
Percentage bioavailability | 192.81 [162.47 to 228.80] | 539.66 [454.37 to 640.96] | 279.90 [235.86 to 332.16]

36. Primary Outcome: Part B: Frel of GSK2982772 Based on AUC (0-24) for MR Coated Tablet Formulation in Fasted State
Description: Blood samples were collected at indicated time points for analysis of Frel (dose) based on AUC(0-24) of GSK2982772. Frel (dose) for AUC(0-24) was calculated as Geometric mean of AUC(0-24) of MR formulation (test dose) Fasted/Geometric mean of AUC(0-24) of MR Fasted formulation (reference dose) multiplied by 100.
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, and 24 hours post-dose
Population: PK Population.
Measure: Number (90% Confidence Interval); unit: Percentage bioavailability
Arm/Group | Part B: MR-16h 960mg Fasted vs MR-16h 480mg Fasted | Part B: MR-16h 960mg Fasted vs MR-16h 120mg Fasted | Part B: MR-16h 480mg Fasted vs MR-16h 120mg Fasted
Number analyzed (Participants) | 16 | 15 | 16
Percentage bioavailability | 175.58 [143.34 to 215.08] | 392.65 [320.16 to 481.54] | 223.63 [182.56 to 273.93]

37. Primary Outcome: Part B: Frel of GSK2982772 Based on Cmax for MR Coated Tablet Formulation in Fasted State
Description: Blood samples were collected at indicated time points for analysis of Frel dose. Frel for Cmax was calculated as Geometric mean of Cmax of MR formulation (test) Fasted/ Geometric mean of Cmax of MR Fasted Formulation (reference dose) multiplied by 100.
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 36 and 48 hours post-dose
Population: PK Population.
Measure: Number (90% Confidence Interval); unit: Percentage bioavailability
Arm/Group | Part B: MR-16h 960mg Fasted vs MR-16h 480mg Fasted | Part B: MR-16h 960mg Fasted vs MR-16h 120mg Fasted | Part B: MR-16h 480mg Fasted vs MR-16h 120mg Fasted
Number analyzed (Participants) | 16 | 15 | 16
Percentage bioavailability | 160.00 [128.12 to 199.81] | 338.70 [270.88 to 423.89] | 211.68 [169.51 to 264.35]

38. Primary Outcome: Part A: Relative Bioavailability (Frelformulation) Based on AUC (0-inf) of GSK2982772 240 mg
Description: Blood samples were collected at indicated time points for analysis of Frelformulation based on AUC(0-inf) of GSK2982772 in fasted state. Frel for AUC(0-inf) was calculated as Geometric mean of AUC(0-inf) of MR formulation (test) Fasted/ Geometric mean of AUC(0-inf) of Fasted of IR Formulation (reference) multiplied by 100.
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 36 and 48 hours post-dose
Population: PK Population.
Measure: Number (90% Confidence Interval); unit: Percentage bioavailability
Groups:
- Part A: MR-12h 240mg Fasted and IR 240mg Fasted: Participants received a single oral dose of 240 mg GSK2982772 MR-12h (80% release in 12 hours) tablet in fasted state and received a single oral dose of 240 mg GSK2982772 IR tablet in fasted state
- Part A: MR-16h 240mg Fasted and IR 240mg Fasted: Participants received a single oral dose of 240 mg GSK2982772 MR-16h (80% release in 16 hours) tablet in fasted state and received a single oral dsoe of 240 mg GSK2982772 IR tablet in fasted state
- Part A: MR-18h 240mg Fasted and IR 240mg Fasted: Participants received a single oral dose of 240 mg GSK2982772 MR-18h (80% release in 18 hours) tablet in fasted state and received a single oral dose of 240 mg GSK2982772 IR tablet in fasted state
Arm/Group | Part A: MR-12h 240mg Fasted and IR 240mg Fasted | Part A: MR-16h 240mg Fasted and IR 240mg Fasted | Part A: MR-18h 240mg Fasted and IR 240mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
Percentage bioavailability | 54.68 [47.64 to 62.76] | 48.32 [40.96 to 57.01] | 57.69 [50.58 to 65.80]

39. Primary Outcome: Part A: Frelformulation Based on AUC (0-t) of GSK2982772 for MR Coated Tablet Formulation (240 mg)
Description: Blood samples were collected at indicated time points for analysis of Frelformulation based on AUC of GSK2982772 in fasted state. Frel for AUC (0-t) was calculated as Geometric mean of AUC(0-t) of MR Fasted formulation (test) / Geometric mean of AUC(0-t) of Fasted of IR Formulation (reference) multiplied by 100.
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 36 and 48 hours
Population: PK Population.
Measure: Number (90% Confidence Interval); unit: Percentage bioavailability
Arm/Group | Part A: MR-12h 240mg Fasted and IR 240mg Fasted | Part A: MR-16h 240mg Fasted and IR 240mg Fasted | Part A: MR-18h 240mg Fasted and IR 240mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
Percentage bioavailability | 57.72 [51.51 to 64.69] | 49.61 [43.86 to 56.11] | 54.86 [49.03 to 61.39]

40. Primary Outcome: Part A: Frelformulation Based on AUC(0-24) of GSK2982772 for MR Coated Tablet Formulation (240 mg)
Description: Blood samples were collected at indicated time points for analysis of Frelformulation based on AUC of GSK2982772 in fasted state. Frel for AUC(0-24) was calculated as Geometric mean of AUC(0-24) of MR Fasted formulation (test) / Geometric mean of AUC(0-24) of Fasted of IR Formulation (reference) multiplied by 100.
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, and 24 hours
Population: PK Population.
Measure: Number (90% Confidence Interval); unit: Percentage bioavailability
Arm/Group | Part A: MR-12h 240mg Fasted and IR 240mg Fasted | Part A: MR-16h 240mg Fasted and IR 240mg Fasted | Part A: MR-18h 240mg Fasted and IR 240mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
Percentage bioavailability | 47.77 [41.92 to 54.43] | 36.85 [31.99 to 42.45] | 40.54 [35.63 to 46.13]

41. Primary Outcome: Part A: Frelformulation Based on Cmax of GSK2982772 for MR Coated Tablet Formulation (240 mg)
Description: Blood samples were collected at indicated time points for analysis of Frelformulation based on Cmax of GSK2982772 in fasted state. Frel for Cmax was calculated as Geometric mean of Cmax of MR Fasted formulation (test) / Geometric mean of Cmax of Fasted Formulation of IR formulation (reference) multiplied by 100.
Time Frame: Pre-dose, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 36 and 48 hours
Population: PK Population.
Measure: Number (90% Confidence Interval); unit: Percentage bioavailability
Arm/Group | Part A: MR-12h 240mg Fasted and IR 240mg Fasted | Part A: MR-16h 240mg Fasted and IR 240mg Fasted | Part A: MR-18h 240mg Fasted and IR 240mg Fasted
Number analyzed (Participants) | 16 | 16 | 16
Percentage bioavailability | 22.29 [18.77 to 26.47] | 14.16 [11.75 to 17.06] | 16.58 [13.99 to 19.66]

42. Secondary Outcome: Part A: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participants, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is defined as any untoward medical occurrence that at any dose may result in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly or birth defect and important medical events that may jeopardize the participants or may require medical or surgical intervention to prevent one of the other outcomes listed before.
Time Frame: Up to Day 67
Population: Safety Population consisted of all participants who receive at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: IR 240 mg Fasted | Part A: MR-12h 240 mg Fasted | Part A: MR-18h 240 mg Fasted | Part A: MR-12h 240 mg Fed (High-Fat) | Part A: MR-18h 240 mg Fed (High-fat) | Part A: MR-16h 240 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16 | 12 | 16 | 12
Participants
  Any AEs | 2 | 5 | 3 | 3 | 3 | 4
  Any SAEs | 0 | 0 | 0 | 0 | 0 | 0

43. Secondary Outcome: Part A: Number of Participants With Emergent Clinical Chemistry Results by Potential Clinical Importance (PCI) Criteria
Description: Clinical chemistry parameters with PCI values:albumin (low: <30 millimoles per liter[mmol/L]), Alanine transaminase (ALT) (high: >=2xupper limit of normal [ULN]), Aspartate Aminotransferase(AST) (high: >=2xULN), Alkaline phosphatase(ALP) (high:>=2xULN), calcium(low: <2 mmol/L, high: >2.75 mmol/L),creatinine (high: >44.2 mmol/L),glucose (low: <3 mmol/L,high: >9 mmol/L), potassium (low: <3 mmol/L,high: >5.5 mmol/L),sodium (low: <130 mmol/L,high: >150 mmol/L),total bilirubin(high :>= 1.5xULN). Participants are counted in the worst case category that their value changes to (Low, Normal or High), unless there is no change in their category. Participants whose value category was unchanged (e.g., High to High),or whose value became normal, are recorded in the "To Normal or No Change" category. Participants are counted twice if the participants has values that changed 'To Low' and 'To High', so the percentages may not add to 100%. Data for worst-case post-Baseline has been reported.
Time Frame: Up to Day 67
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: IR 240 mg Fasted | Part A: MR-12h 240 mg Fasted | Part A: MR-18h 240 mg Fasted | Part A: MR-12h 240 mg Fed (High-Fat) | Part A: MR-18h 240 mg Fed (High-fat) | Part A: MR-16h 240 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16 | 12 | 16 | 12
Participants
  ALT, To Normal or No Change | 16 | 16 | 16 | 12 | 16 | 12
  ALT, To High | 0 | 0 | 0 | 0 | 0 | 0
  AST, To Normal or No Change | 16 | 16 | 16 | 12 | 16 | 12
  AST, To High | 0 | 0 | 0 | 0 | 0 | 0
  ALP, To Normal or No Change | 16 | 16 | 16 | 12 | 16 | 12
  ALP, To High | 0 | 0 | 0 | 0 | 0 | 0
  Albumin, To low | 0 | 0 | 0 | 0 | 0 | 0
  Albumin, To Normal or no Change | 16 | 16 | 16 | 12 | 16 | 12
  Calcium, To low | 0 | 0 | 0 | 0 | 2 | 0
  Calcium, To Normal or No Change | 16 | 16 | 16 | 12 | 14 | 12
  Calcium, To High | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine, To Normal or No Change | 16 | 16 | 16 | 12 | 16 | 12
  Creatinine, To High | 0 | 0 | 0 | 0 | 0 | 0
  Glucose, To low | 0 | 0 | 0 | 0 | 0 | 0
  Glucose, To Normal or No Change | 16 | 16 | 16 | 12 | 16 | 12
  Glucose, To High | 0 | 0 | 0 | 0 | 0 | 0
  Potassium, To low | 0 | 0 | 0 | 0 | 0 | 0
  Potassium, To Normal or No Change | 16 | 16 | 16 | 12 | 16 | 12
  Potassium, To High | 0 | 0 | 0 | 0 | 0 | 0
  Sodium, To low | 0 | 0 | 0 | 0 | 0 | 0
  Sodium, To Normal or No Change | 16 | 16 | 16 | 12 | 16 | 12
  Sodium, To High | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin, To Normal or No Change | 16 | 16 | 16 | 12 | 16 | 12
  Total Bilirubin, To High | 0 | 0 | 0 | 0 | 0 | 0

44. Secondary Outcome: Part A: Number of Participants With Emergent Hematology Results by Potential Clinical Importance Criteria
Description: Hematology parameters with PCI ranges: hematocrit (high: >0.54 percentage of red blood cells), hemoglobin (high: >180 grams per liter [g/L]), lymphocytes (low: <0.8*giga cells per liter [10^9/L]), total neutrophil count (low: <1.5*10^9/L), platelet count (low: <100*10^9/L and high: >550*10^9/L), and while blood cell (WBC) count (low: <3*10^9/L and high: >20*10^9/L). Participants are counted in the worst case category that their value changes to (Low, Normal or High), unless there is no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became normal, are recorded in the "To Normal or No Change" category. Participants are counted twice if the subject has values that changed 'To Low' and 'To High', so the percentages may not add to 100%. Data for worst-case post-Baseline has been reported.
Time Frame: Up to Day 67
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: IR 240 mg Fasted | Part A: MR-12h 240 mg Fasted | Part A: MR-18h 240 mg Fasted | Part A: MR-12h 240 mg Fed (High-Fat) | Part A: MR-18h 240 mg Fed (High-fat) | Part A: MR-16h 240 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16 | 12 | 16 | 12
Participants
  Hemotocrit, To Normal or No Change | 16 | 16 | 16 | 12 | 16 | 12
  Hematocrit, To High | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin, To Normal or No Change | 16 | 16 | 16 | 12 | 16 | 12
  Hemoglobin, To High | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes, To Low | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes, To Normal or No Change | 16 | 16 | 16 | 12 | 16 | 12
  Platelet count, To Low | 0 | 0 | 0 | 0 | 0 | 0
  Platelet count, To Normal or No change | 16 | 16 | 16 | 12 | 16 | 12
  Platelet count, To High | 0 | 0 | 0 | 0 | 0 | 0
  Total neutrophils, To Low | 0 | 0 | 0 | 0 | 0 | 0
  Total Neutrophils, To Normal or No Change | 16 | 16 | 16 | 12 | 16 | 12
  WBC count, To Low | 0 | 0 | 0 | 0 | 0 | 0
  WBC count, To Normal or no Change | 16 | 16 | 16 | 12 | 16 | 12
  WBC count, To High | 0 | 0 | 0 | 0 | 0 | 0

45. Secondary Outcome: Part A: Number of Participants With Abnormal Urinalysis Dipstick Results
Description: Urine samples were collected for analysis of specific gravity, potential of hydrogen ions, glucose, protein, blood and ketones by dipstick method. Microscopic examination was performed abnormal data for red blood cells (RBC): 1-9 High potential field (HPF) and WBC: 1-9/ HPF; WBC: 10-50/HPF has been presented.
Time Frame: Day 2 (post-dose)
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: IR 240 mg Fasted | Part A: MR-12h 240 mg Fasted | Part A: MR-18h 240 mg Fasted | Part A: MR-12h 240 mg Fed (High-Fat) | Part A: MR-18h 240 mg Fed (High-fat) | Part A: MR-16h 240 mg Fasted
Number analyzed (Participants) | 16 | 16 | 16 | 12 | 16 | 12
Participants
  RBC 1-9/ HPF | 0 | 2 | 0 | 1 | 0 | 0
  WBC 1-9/HPF | 1 | 1 | 1 | 4 | 1 | 3
  WBC 10-50/HPF | 2 | 0 | 1 | 0 | 0 | 0

46. Secondary Outcome: Part A: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) in IR Formulation
Description: SBP and DBP were measured in a semi-supine position after 5 minutes of rest of the participant. Baseline is defined as the latest pre-dose assessment before entering study. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Day 1: 2 and 12 hours; Day 2: 24 hours
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part A: IR 240 mg Fasted
Number analyzed (Participants) | 16
Millimeters of mercury
  SBP, Day 1, 2 hours | -3.9 (6.29)
  SBP, Day 1, 12 hours | -3.3 (6.39)
  SBP, Day 2, 24 hours | -6.6 (7.26)
  DBP, Day1, 2 hours | -1.1 (3.00)
  DBP, Day 1, 12 hours | -5.1 (3.51)
  DBP, Day 2, 24 hours | -1.4 (4.63)

47. Secondary Outcome: Part A: Change From Baseline in SBP and DBP in MR Formulation
Description: as for outcome 46
Time Frame: Baseline (Day 1, Pre-dose), Day 1: 2 and 12 hours; Day 2: 24 hours, Day 3: 48 hours
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part A: MR-12h 240 mg Fasted | Part A: MR-18h 240 mg Fasted | Part A: MR-12h 240 mg Fed (High-Fat) | Part A: MR-18h 240 mg Fed (High-fat) | Part A: MR-16h 240 mg Fasted
Number analyzed (Participants) | 16 | 16 | 12 | 16 | 12
Millimeters of mercury
  SBP, Day1, 2 hours | -2.7 (5.76) | -7.9 (6.82) | -7.3 (8.57) | -4.6 (8.38) | -3.4 (9.18)
  SBP, Day1, 12 hours | -3.0 (8.07) | -6.9 (8.32) | -2.4 (10.07) | -0.09 (13.02) | -1.3 (10.54)
  SBP, Day 2, 24 hours | -3.9 (7.55) | -10.3 (8.69) | -2.8 (8.87) | -6.8 (5.72) | -2.3 (7.01)
  SBP, Day3, 48 hours, | -2.0 (9.29) | -5.3 (7.15) | -1.7 (8.87) | -4.2 (7.74) | 2.8 (7.88)
  DBP, Day1, 2 hours | -4.5 (5.67) | -5.3 (5.70) | -6.1 (3.53) | -6.9 (5.11) | -2.3 (8.64)
  DBP, Day1, 12 hours | -7.6 (7.46) | -8.3 (5.35) | -5.7 (5.14) | -5.9 (6.35) | -5.3 (7.12)
  DBP, Day2, 24 hours | -2.4 (6.30) | -10.0 (4.15) | -6.6 (5.76) | -4.5 (4.93) | -0.4 (6.82)
  DBP, Day3, 48 hours | -3.7 (6.26) | -3.7 (4.71) | -2.1 (7.33) | -2.4 (5.20) | -1.1 (7.74)

48. Secondary Outcome: Part A: Change From Baseline in Heart Rate in IR Formulation
Description: Heart rate was measured in a semi-supine position after 5 minutes of rest of participant. Baseline is defined as the latest pre-dose assessment before entering study. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Day 1: 2 and 12 hours; Day 2: 24 hours
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part A: IR 240 mg Fasted
Number analyzed (Participants) | 16
Beats per minute
  Day 1, 2 hours | -2.6 (8.37)
  Day 1, 12 hours | 6.3 (11.51)
  Day 2, 24 hours | -2.1 (7.73)

49. Secondary Outcome: Part A: Change From Baseline in Heart Rate in MR Formulation
Description: as for outcome 48
Time Frame: Baseline (Day 1, Pre-dose), Day 1: 2 and 12 hours; Day 2: 24 hours, Day 3: 48 hours
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part A: MR-12h 240 mg Fasted | Part A: MR-18h 240 mg Fasted | Part A: MR-12h 240 mg Fed (High-Fat) | Part A: MR-18h 240 mg Fed (High-fat) | Part A: MR-16h 240 mg Fasted
Number analyzed (Participants) | 16 | 16 | 12 | 16 | 12
Beats per minute
  Day 1, 2 hours | -1.3 (7.22) | -6.1 (7.78) | 5.8 (6.87) | 3.1 (7.33) | -1.3 (5.87)
  Day 1, 12 hours | 5.4 (9.62) | 6.1 (9.79) | 9.8 (7.72) | 3.4 (10.19) | 8.8 (8.41)
  Day 2, 24 hours | 0.7 (7.36) | -4.7 (8.72) | 2.4 (8.56) | 1.6 (9.21) | -2.4 (4.12)
  Day 3, 48 hours | 8.6 (11.39) | 0.4 (8.58) | 3.8 (5.67) | 4.7 (9.71) | 7.3 (7.19)

50. Secondary Outcome: Part A: Change From Baseline in Respiration Rate in IR Formulation
Description: Respiratory rate was measured in a semi-supine position after 5 minutes of rest of the participant. Baseline is defined as the latest pre-dose assessment before entering study. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Day 1: 2 and 12 hours; Day 2: 24 hours
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part A: IR 240 mg Fasted
Number analyzed (Participants) | 16
Breaths per minute
  Day 1, 2 hours | -0.4 (3.08)
  Day 1, 12 hours | -0.2 (2.10)
  Day 2, 24 hours | -0.8 (3.53)

51. Secondary Outcome: Part A: Change From Baseline in Respiration Rate in MR Formulation
Description: as for outcome 50
Time Frame: Baseline (Day 1, Pre-dose), Day 1: 2 and 12 hours; Day 2: 24 hours, Day 3: 48 hours
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part A: MR-12h 240 mg Fasted | Part A: MR-18h 240 mg Fasted | Part A: MR-12h 240 mg Fed (High-Fat) | Part A: MR-18h 240 mg Fed (High-fat) | Part A: MR-16h 240 mg Fasted
Number analyzed (Participants) | 16 | 16 | 12 | 16 | 12
Breaths per minute
  Day 1, 2 hours; n=16, 16, 12, 16, 12 | 0.9 (2.89) | 2.5 (2.58) | 2.8 (2.29) | 2.0 (2.13) | 0.0 (3.25)
  Day 1, 12 hours; n=15, 16, 12, 16, 12: number analyzed (Participants) | 15 | 16 | 12 | 16 | 12
  Day 1, 12 hours; n=15, 16, 12, 16, 12 | 1.1 (1.68) | 0.8 (1.94) | 2.2 (2.25) | 0.9 (2.14) | 2.1 (3.34)
  Day 2, 24 hours; n=16, 16, 12, 16, 12 | 1.4 (1.93) | 0.9 (2.58) | 1.9 (2.43) | 2.2 (1.64) | 0.9 (2.68)
  Day 3, 48 hours; n=16, 16, 12, 16, 12 | 2.3 (3.00) | 0.4 (1.79) | 4.0 (2.37) | 0.7 (1.99) | -0.4 (2.64)

52. Secondary Outcome: Part A: Change From Baseline in Body Temperature in IR Formulation
Description: Body temperature was measured in semi-supine position. Baseline is defined as the latest pre-dose assessment before entering study. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Day 1: 2 and 12 hours; Day 2: 24 hours
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Part A: IR 240 mg Fasted
Number analyzed (Participants) | 16
Degrees Celsius
  Day 1, 2 hours | 0.04 (0.159)
  Day 1, 12 hours | 0.13 (0.241)
  Day 2, 24 hours | 0.10 (0.183)

53. Secondary Outcome: Part A: Change From Baseline in Body Temperature in MR Formulation
Description: as for outcome 52
Time Frame: Baseline (Day 1, Pre-dose), Day 1: 2 and 12 hours; Day 2: 24 hours, Day 3: 48 hours
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Part A: MR-12h 240 mg Fasted | Part A: MR-18h 240 mg Fasted | Part A: MR-12h 240 mg Fed (High-Fat) | Part A: MR-18h 240 mg Fed (High-fat) | Part A: MR-16h 240 mg Fasted
Number analyzed (Participants) | 16 | 16 | 12 | 16 | 12
Degrees Celsius
  Day 1, 2 hours | -0.04 (0.216) | 0.14 (0.190) | -0.03 (0.107) | -0.06 (0.141) | -0.04 (0.211)
  Day 1, 12 hours | 0.12 (0.180) | 0.15 (0.266) | 0.11 (0.162) | -0.04 (0.150) | 0.24 (0.188)
  Day 2, 24 hours | -0.03 (0.188) | 0.12 (0.148) | 0.06 (0.151) | 0.05 (0.175) | 0.08 (0.175)
  Day 3, 48 hours | -0.05 (0.163) | 0.01 (0.247) | 0.04 (0.156) | 0.01 (0.178) | 0.07 (0.222)

54. Secondary Outcome: Part A: Number of Participants With Abnormal Electrocardiogram (ECG) Findings in IR Formulation
Description: Single 12-lead ECGs were obtained using an automated ECG machine that calculated PR, QRS, QT and Corrected QT (QTc) intervals. ECG measurements were performed in a semi-supine or supine position. Number of participants with abnormal clinically significant findings and abnormal not clinically significant findings in ECG results has been reported. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Data for worst-case post-Baseline has been reported.
Time Frame: Up to Day 67
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: IR 240 mg Fasted
Number analyzed (Participants) | 16
Participants
  Abnormal-Not Clinically Significant | 8
  Abnormal - Clinically Significant | 0

55. Secondary Outcome: Part A: Number of Participants With Abnormal Electrocardiogram (ECG) Findings in MR Formulation
Description: as for outcome 54
Time Frame: Up to Day 67
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: MR-12h 240 mg Fasted | Part A: MR-18h 240 mg Fasted | Part A: MR-12h 240 mg Fed (High-Fat) | Part A: MR-18h 240 mg Fed (High-fat) | Part A: MR-16h 240 mg Fasted
Number analyzed (Participants) | 16 | 16 | 12 | 16 | 12
Participants
  Abnormal-Not Clinically Significant | 8 | 10 | 5 | 9 | 7
  Abnormal - Clinically Significant | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Non-serious AEs and SAEs were collected up to Day 67 for Part A and up to Day 68 for Part B
Description: Non-serious AEs and SAEs were collected in Safety population.
Groups:
- Part A: MR-18h 240mg Fasted: Participants received a single oral dose of 240 mg GSK2982772 MR-18h tablet in fasted state
- Part A: MR-18h 240mg Fed (High-Fat): Participants received a single oral dose of 240 mg GSK2982772 MR-18h tablet after high fat meal in fed state
- Part A: MR-16h 240mg Fasted: Participants received a single oral dose of 240 mg GSK2982772 MR-16h tablet in fasted state
- Part B: MR-16h 480mg Fasted: Participants received a single oral dose of 480 mg GSK2982772 MR-16 h (80% release in 16 hours) tablet in fasted state
- Part B: MR-16h 480 mg Fed (Std): Participants received a single oral dose of 480 mg GSK2982772 MR-16h (80% release in 16 hours) tablet after a standard breakfast (fed state)
- Part B: MR-16h 960mg Fasted: Participants received a single oral dose of 960 mg GSK2982772 MR-16h (80% release in 16 hours) tablet in fasted state
- Part B: MR-16h 120mg Fasted: Participants received 120 mg GSK2982772 MR-16 h (80% release in 16 hours) tablet in fasted state
Arm/Group | Part A: IR 240 mg Fasted | Part A: MR-12h 240 mg Fasted | Part A: MR-18h 240mg Fasted | Part A: MR-12h 240mg Fed (High-Fat) | Part A: MR-18h 240mg Fed (High-Fat) | Part A: MR-16h 240mg Fasted | Part B: MR-16h 480mg Fasted | Part B: MR-16h 480 mg Fed (Std) | Part B: MR-16h 480mg Fed (High-fat) | Part B: MR-16h 480mg Fed (High-Fat) (Enteric Coated) | Part B: MR-16h 960mg Fasted | Part B: MR-16h 120mg Fasted
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/12 | 0/16 | 0/12 | 0/16 | 0/14 | 0/15 | 0/14 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/12 | 0/16 | 0/12 | 0/16 | 0/14 | 0/15 | 0/14 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 2/16 | 5/16 | 3/16 | 3/12 | 3/16 | 4/12 | 8/16 | 4/14 | 1/15 | 3/14 | 3/15 | 3/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: IR 240 mg Fasted (N=16) | Part A: MR-12h 240 mg Fasted (N=16) | Part A: MR-18h 240mg Fasted (N=16) | Part A: MR-12h 240mg Fed (High-Fat) (N=12) | Part A: MR-18h 240mg Fed (High-Fat) (N=16) | Part A: MR-16h 240mg Fasted (N=12) | Part B: MR-16h 480mg Fasted (N=16) | Part B: MR-16h 480 mg Fed (Std) (N=14) | Part B: MR-16h 480mg Fed (High-fat) (N=15) | Part B: MR-16h 480mg Fed (High-Fat) (Enteric Coated) (N=14) | Part B: MR-16h 960mg Fasted (N=15) | Part B: MR-16h 120mg Fasted (N=15)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Application site irritation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT03649412/SAP_000.pdf
  • Study Protocol (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT03649412/Prot_001.pdf